CLINICAL TRIAL: NCT06045221
Title: A Phase 3, Randomized, Open-Label Study to Investigate the Efficacy and Safety of Once Daily Oral LY3502970 Compared With Oral Semaglutide in Adult Participants With Type 2 Diabetes and Inadequate Glycemic Control With Metformin (ACHIEVE-3)
Brief Title: A Study of Orforglipron (LY3502970) Compared With Semaglutide in Participants With Type 2 Diabetes Inadequately Controlled With Metformin
Acronym: ACHIEVE-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18565; J2A-MC-GZGU (Other: Eli Lilly and Company); U1111-1290-6014 (Other: UTN Number)
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — orforglipron; semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Orforglipron Dose 1 (Experimental): Participants will receive orforglipron orally.
  Interventions: Drug: Orforglipron
- Orforglipron Dose 2 (Experimental): Participants will receive orforglipron orally.
  Interventions: Drug: Orforglipron
- Semaglutide Dose 1 (Active Comparator): Participants will receive semaglutide orally.
  Interventions: Drug: Semaglutide
- Semaglutide Dose 2 (Active Comparator): Participants will receive semaglutide orally.
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Orforglipron — Administered orally
  Other Names: LY3502970
  Arms: Orforglipron Dose 1; Orforglipron Dose 2
Drug: Semaglutide — Administered orally
  Arms: Semaglutide Dose 1; Semaglutide Dose 2

SUMMARY:
The main purpose of this study is to assess efficacy and safety of orforglipron compared with oral semaglutide in participants with Type 2 diabetes and inadequate glycemic control with metformin.The study will last around 61 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have Type 2 Diabetes
* Have HbA1c ≥7.0% (53 mmol/mol) to ≤10.5% (91 mmol/mol), as determined by the central laboratory at screening.
* Have been on stable diabetes treatment with metformin ≥1500 milligram (mg)/day during the 90 days prior to screening and maintained through randomization.
* Are of stable body weight (±5%) for at least 90 days prior to screening and agree to not initiate an intensive diet or exercise program during the study with the intent of reducing body weight, other than the lifestyle and/or dietary measures for diabetes treatment

Exclusion Criteria:

* Have Type 1 Diabetes
* Are currently receiving or planning to receive treatment for diabetic retinopathy and/or macular edema, for example, laser photocoagulation or intravitreal injections of anti-vascular endothelial growth factor inhibitors.
* Have a history of ketoacidosis or hyperosmolar state or coma within the last 6 months prior to screening, or between screening and randomization.
* Have a New York Heart Association functional classification IV congestive heart failure.
* Have an estimated glomerular filtration rate (eGFR) <45 milliliter/minute (mL/min)/1.73 square meter (m²) or lower than the country-specific threshold for discontinuing metformin therapy per local label as determined by the central laboratory at screening.
* Have a serum calcitonin level of ≥35 nanogram/Liter (ng/L), as determined by the central laboratory at screening.
* Have a history of an active or untreated malignancy or are in remission from a clinically significant malignancy for less than 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1698 (Actual)
Dates: Start 2023-09-22 (Actual); Primary Completion 2025-08-22 (Actual); Study Completion 2025-08-22 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Hemoglobin A1c (HbA1c) | Baseline, Week 52

SECONDARY OUTCOMES:
Change from Baseline in HbA1c | Baseline, Week 52
Percentage of Participants Who Achieved HbA1c <7.0% 53 millimole/mole (mmol/mol) | Week 52
Percentage of Participants Who Achieved HbA1c ≤6.5% (48 mmol/mol) | Week 52
Percentage Change from Baseline in Body Weight | Baseline, Week 52
Change from Baseline in Body Weight | Baseline, Week 52
Percentage of Participants Who Achieved HbA1c <5.7% (39 mmol/mol) | Week 52
Change from Baseline in Fasting Serum Glucose | Baseline, Week 52
Change from Baseline in Daily Average 7-point Self-monitored Blood Glucose (SMBG) | Baseline, Week 52
Percentage of Participants Who Achieved Weight Loss of ≥5% | Week 52
Percentage of Participants Who Achieved Weight Loss of ≥10% | Week 52
Percentage of Participants Who Achieved Weight Loss of ≥15% | Week 52
Change from Baseline in Systolic Blood Pressure (SBP) | Baseline, Week 52
Change from Baseline in Diastolic Blood Pressure (DBP) | Baseline, Week 52
Percentage Change from Baseline in Total Cholesterol | Baseline, Week 52
Percentage Change from Baseline in High Density Lipoprotein (HDL)-Cholesterol | Baseline, Week 52
Percentage Change from Baseline in Low Density Lipoprotein (LDL)-Cholesterol | Baseline, Week 52
Percentage Change from Baseline in Very Low Density Lipoprotein (VLDL)-Cholesterol | Baseline, Week 52
Percentage Change from Baseline in Non-HDL-Cholesterol | Baseline, Week 52
Percentage Change from Baseline in Triglycerides | Baseline, Week 52
Change from Baseline in Short Form 36 Version 2 (SF-36-v2) Acute Form Domain Summary Scores | Baseline, Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (131):
- United States (64):
  - Absolute Clinical Research, Phoenix, Arizona
  - San Fernando Valley Health Institute, Canoga Park, California
  - Neighborhood Healthcare Institute of Health, Escondido, California
  - Velocity Clinical Research, Gardena, Gardena, California
  - Biopharma Informatic, LLC, Los Angeles, California
  - Velocity Clinical Research, Westlake, Los Angeles, California
  - Infinity Clinical Research - Norco, Norco, California
  - Valley Clinical Trials, Inc., Northridge, California
  - Norcal Endocrinology & Internal Medicine, San Ramon, California
  - Encompass Clinical Research, Spring Valley, California
  - University Clinical Investigators, Inc., Tustin, California
  - New West Physicians Clinical Research, Golden, Colorado
  - Connecticut Clinical Research - Cromwell, Cromwell, Connecticut
  - Clinical Research of West Florida, Inc. (Clearwater), Clearwater, Florida
  - South Florida Clinical Research Institute, Margate, Florida
  - Miami Dade Medical Research Institute, LLC, Miami, Florida
  - West Orange Endocrinology, Ocoee, Florida
  - Latin Clinical Trial Center Florida, Tamarac, Florida
  - Clinical Research of West Florida, Tampa, Florida
  - Metabolic Research Institute, Inc., West Palm Beach, Florida
  - Balanced Life Health Care Solutions/SKYCRNG, Lawrenceville, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - North Georgia Clinical Research, Woodstock, Georgia
  - Northwest Clinical Trials, Boise, Idaho
  - Family First Medical Center, Idaho Falls, Idaho
  - American Health Network of Indiana, LLC - Greenfield, Greenfield, Indiana
  - Velocity Clinical Research, Valparaiso, Valparaiso, Indiana
  - Cotton O'Neil Diabetes & Endocrinology, Topeka, Kansas
  - Tekton Research, Inc, Wichita, Kansas
  - DelRicht Research, New Orleans, Louisiana
  - Joslin Diabetes Center, Boston, Massachusetts
  - Revival Research Institute, LLC, Dearborn, Michigan
  - SKY Integrative Medical Center/SKYCRNG, Ridgeland, Mississippi
  - Kansas City Research Institute, Kansas City, Missouri
  - Logan Health Research, Kalispell, Montana
  - Wr-Crcn, Llc, Las Vegas, Nevada
  - Premier Research, Trenton, New Jersey
  - Albany Medical College, Division of Community Endocrinology, Albany, New York
  - Ellipsis Research Group - Brooklyn - 7th Street, Brooklyn, New York
  - Great Lakes Medical Research, LLC, Westfield, New York
  - PharmQuest Life Sciences, LLC, Greensboro, North Carolina
  - Lucas Research, Inc, Morehead City, North Carolina
  - Accellacare - Piedmont, Statesville, North Carolina
  - Wake Forest University Baptist Medical Center (WFUBMC), Winston-Salem, North Carolina
  - Aventiv Research Inc, Columbus, Ohio
  - Tekton Research, Inc, Moore, Oklahoma
  - Alliance for Multispecialty Research, LLC, Norman, Oklahoma
  - The Corvallis Clinic, P.C., Corvallis, Oregon
  - Heritage Valley Medical Group, Inc., Beaver, Pennsylvania
  - Preferred Primary Care Physicians, Preferred Clinical Research (Ofc 18), Pittsburgh, Pennsylvania
  - The Research Center of The Upstate, Greenville, South Carolina
  - New Phase Research and Development, Knoxville, Tennessee
  - Clinical Neuroscience Solutions Inc., Memphis, Tennessee
  - Velocity Clinical Research, Austin, Austin, Texas
  - Velocity Clinical Research, Dallas, Dallas, Texas
  - Diabetes and Thyroid Center of Ft. Worth, Fort Worth, Texas
  - Juno Research, Houston, Texas
  - Endocrine Ips, Pllc, Houston, Texas
  - Clear Brook Medical Associates, Houston, Texas
  - Southern Endocrinology Associates, Mesquite, Texas
  - Texas Valley Clinical Research, Weslaco, Texas
  - Synexus Clinical Research US, Inc., Salt Lake City, Utah
  - Eastside Research Associates, Redmond, Washington
  - Rainier Clinical Research Center, Renton, Washington
- Argentina (17):
  - Centro de Investigaciones Metabólicas (CINME), Ciudad Autónoma de Buenos Aires, Buenos Aires
  - CIMeL, Lanús, Buenos Aires
  - Centro de Investigaciones Médicas Mar del Plata, Mar del Plata, Buenos Aires
  - Policlinica Red OMIP, Mar del Plata, Buenos Aires
  - Consultorio de Investigación Clínica EMO SRL, Buenos Aires, Buenos Aires F.D.
  - CIPREC, Buenos Aires, Buenos Aires F.D.
  - Centro Médico Viamonte, Buenos Aires, Buenos Aires F.D.
  - Instituto Centenario, CABA, Buenos Aires F.D.
  - Centro de Salud e Investigaciones Médicas, Santa Rosa, La Pampa Province
  - INECO Neurociencias Oroño, Rosario, Santa Fe Province
  - Instituto de Especialidades de la Salud Rosario, Rosario, Santa Fe Province
  - Instituto Médico Catamarca IMEC, Rosario, Santa Fe Province
  - Instituto Médico Fundación Grupo Colaborativo Rosario Investigación y Prevención Medica, Rosario, Santa Fe Province
  - Fundacion Estudios Clinicos, Rosario, Santa Fe Province
  - Instituto de Investigaciones Clínicas Córdoba, Córdoba
  - Instituto Médico DAMIC, Córdoba
  - Sanatorio Norte, Santiago del Estero
- China (21):
  - Beijing Pinggu District Hospital, Beijing, Beijing Municipality
  - Chongqing General Hospital, Chongqing, Chongqing Municipality
  - Shunde Hospital of Southern Medical Univesity, Foshan, Guangdong
  - Huizhou Municipal Central Hospital, Huizhou, Guangdong
  - The Fourth Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang Shi, Henan
  - Nanyang First People's Hospital, Nanyang, Henan
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Nanjing First Hospital, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - Jiangxi Pingxiang People's Hospital, Pingxiang, Jiangxi
  - Dalian Municipal Central Hospital Affiliated of Dalian Medical University, Dalian, Liaoning
  - Jinan Central Hospital, Jinan, Shandong
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - Pudong New Area People's Hospital Shanghai, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Zhejiang Hospital, Hangzhou, Zhejiang
  - Huzhou Central Hospital, Huzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
- Japan (9):
  - Mikannohana Clinic, Diabetes, Endocrinology and Metabolism, Matsuyama, Ehime
  - Manda Memorial Hospital, Sapporo, Hokkaido
  - Nakamoto Internal Medicine Clinic, Mito, Ibaraki
  - Nakakinen clinic, Naka, Ibaraki
  - Ohishi Internal Medicine Clinic, Tsuchiura, Ibaraki
  - Takai Internal Medicine Clinic, Kamakura-shi, Kanagawa
  - Shiraiwa Medical Clinic, Kashihara, Osaka
  - Medical Corporation Sato Medical clinic, Ootaku, Tokyo
  - Gifu University Hospital, Gifu
- Mexico (16):
  - Centro de Investigacion Medica Integral, Guadalajara, Jalisco
  - Instituto Jalisciense de Investigacion en Diabetes y Obesidad, Guadalajara, Jalisco
  - CICEJ Centro de Investigación Clínica Endocrinológica de Jalisco S.C, Guadalajara, Jalisco
  - Private Practice - Dr. Arechavaleta Granell Maria del Rosario, Guadalajara, Jalisco
  - Virgen Cardiovascular Research SC, Guadalajara, Jalisco
  - Centro de Investigacion Medica de Occidente, S.C., Zapopan, Jalisco
  - Caimed Investigacion En Salud S.A. de C.V., Mexico City, Mexico City
  - Centro Especializado En Diabetes, Obesidad Y Prevencion De Enfermedades Cardiovasculares, Mexico City, Mexico City
  - Cardiolink Clin Trials, Monterrey, Nuevo León
  - Unidad biomedica avanzada monterrey, Monterrey, Nuevo León
  - Clínica García Flores SC, Monterrey, Nuevo León
  - Eukarya PharmaSite, Monterrey, Nuevo León
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey, Nuevo León
  - Centro de investigación y control metabólico, San Nicolás de los Garza, Nuevo León
  - Centro Para El Desarrollo de La Medicina Y de Asistencia Medica Especializada S.C., Culiacán, Sinaloa
  - Lahoja. Asociacion Para La Investigacion Y La Farmacovigilancia, Durango
- Puerto Rico (4):
  - Isis Clinical Research Center, Guaynabo, PR
  - Mgcendo Llc, San Juan, PR
  - Research and Cardiovascular Corp., Ponce
  - Latin Clinical Trial Center, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: A Study of Orforglipron (LY3502970) Compared With Semaglutide in Participants With Type 2 Diabetes Inadequately Controlled With Metformin (ACHIEVE-3) — https://trials.lilly.com/en-US/trial/424335